CLINICAL TRIAL: NCT06874335
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation, Dose Expansion and Dose Confirmation Study of BHV-1530 in Adult Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1 Study of BHV-1530 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BHV1530-101
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
Keywords: FGFR3-targeting ADC; antibody-drug conjugate; FGRF3; ADC; FGFR3 alteration; advanced cancers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BHV-1530 Monotherapy (Experimental)
  Interventions: Drug: BHV-1530

INTERVENTIONS:
Drug: BHV-1530 — BHV-1530 will be administered as an IV infusion on Day 1 of each 21-day cycle
  Other Names: AMB302

SUMMARY:
This is a Phase 1, first in human (FIH), open-label, multicenter study of BHV-1530 in adult participants with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written Independent Ethics Committee (IEC)/Institutional Review Board (IRB)-approved informed consent
2. Age greater than or equal to 18 years
3. Participants consent to provide tumor tissue collected prior to study treatment, preferably from a biopsy performed after their last anticancer therapy and within 90 days of the start of study treatment. An older archival sample may be acceptable with Sponsor approval.
4. Participants must have progressed following, are intolerant of, or have no available standard-of-care therapy.
5. Patients with histologically or cytologically confirmed locally advanced/metastatic relapsed or refractory solid tumors as outlined below:

   * Dose-escalation and Dose-expansion (Backfill) Cohorts:

     * Participants with urothelial cancer of the urinary tract: (including renal pelvis, ureters, urinary bladder, and urethra), non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC) regardless of the presence of an activating FGFR3 alteration (mutation, fusion, or amplification) or high FGFR3 protein or mRNA expression in the absence of a detectable genetic alteration.
     * Other advanced or metastatic solid tumors with a documented activating FGFR3 alteration (mutation, fusion, or amplification) or high FGFR3 protein or mRNA expression in the absence of a detectable genetic alteration.
   * Dose Confirmation Cohort:

     * Participants with urothelial cancer of the urinary tract: (including renal pelvis, ureters, urinary bladder, and urethra), non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC) regardless of the presence of an activating FGFR3 alteration (mutation, fusion, or amplification) or high FGFR3 protein or mRNA expression in the absence of a detectable genetic alteration.
     * Other advanced or metastatic solid tumors with a documented activating FGFR3 alteration (mutation, fusion, or amplification) or high FGFR3 protein or mRNA expression in the absence of a detectable genetic alteration, as determined by a validated assay performed in a CLIA certified local or central laboratory.
6. Measurable advanced or metastatic tumors per RECIST 1.1 criteria
7. Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Acceptable liver function:

   * Bilirubin ≤ 1.5 × upper limit of normal (ULN). Participants with known Gilbert's syndrome who have total bilirubin level ≤3×ULN may be enrolled.
   * AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN (if liver metastases are present, then ≤ 5 × ULN is allowed)
9. Acceptable renal function:

   • Serum creatinine ≤1.5 × ULN, or creatinine clearance ≥50 mL/min as calculated using the modified Cockcroft-Gault equation; confirmation of creatinine clearance is only required when creatinine is >1.5 × ULN; 24-hour urine collection is allowed, but not required
10. Acceptable hematologic status:

    * Blood transfusion or growth factor support is not allowed within 7 days prior to blood samples that will be used to establish eligibility
    * Absolute neutrophil count greater than or equal to 1500/mm3. Participants with known Duffy null phenotype who have absolute neutrophil count ≥ 1,200/mm3 may be enrolled
    * Platelet count greater than or equal to 100,000 mm3
    * Hemoglobin greater than or equal to 9 g/dL
    * Activated partial thromboplastin time (aPTT) ≤1.5×ULN. Study participants on therapeutic doses of anticoagulation medication must have INR and/or aPTT ≤ the upper limit of the therapeutic range for intended use
11. A negative urine or serum pregnancy test (if a woman of childbearing potential);
12. Women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and for 7 months (for women) or 4 months (for men) after the last dose of study drug.

Exclusion Criteria:

1. Prior treatment with antibody drug conjugate (ADC) with a topoisomerase-I inhibitor payload. Prior direct treatment with topoisomerase inhibitor (e.g., irinotecan, topotecan, belotecan, nano-liposomal irinotecan) are not exclusionary.
2. Participant has clinically significant intercurrent disease including, but not limited to:

   * New York Heart Association Class III or IV heart failure
   * Myocardial infarction, unstable angina, or stroke ≤ 6 months prior to C1D1
   * Newly diagnosed thromboembolic events that require therapeutic intervention over the last 6 months prior to C1D1 (participants with stable control of lower limb deep venous thrombosis over at least 3 months are allowed)
   * Severe aortic stenosis
   * Uncontrolled arrhythmia
   * Symptomatic pericardial effusion
   * Congenital long QT syndrome
   * A mean of Fredericia's formula-QT corrected interval (QTcF) prolongation to >470 msec based on a 12-lead ECG
   * Uncontrolled hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg) or diabetes (hemoglobin A1C ≥9.0%)
   * Left ventricular ejection fraction (LVEF) <45% determined by echocardiogram or multiple gated acquisition scan (MUGA)
   * Symptomatic pleural effusion (<90% oxygen saturation)
3. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
4. Primary central nervous system (CNS) tumors, current or previously treated leptomeningeal disease or known active brain metastases.

   NOTE: Participants with previously treated, clinically stable, radiologically stable brain metastases maybe eligible
5. Pregnant or nursing women
6. Any standard cancer therapy (e.g., chemotherapy, hormonal therapy, radiotherapy, immunotherapy, biologic therapy treatment) or experimental therapy within 4 weeks or 5 half-lives, whichever is shorter, prior to C1D1. The interval may be reduced to 2 weeks for bone-only radiation therapy. Any major surgical procedure within 6 weeks prior to C1D1
7. Participants have not recovered (i.e., improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia and vitiligo. If the participant has an ongoing, stable, chronic Grade 2 toxicity they may be eligible after discussion with Sponsor on a case-by-case basis
8. Any clinically significant corneal or retinal abnormality that may increase the risk of eye toxicity
9. Known active infection with human immunodeficiency virus (HIV), human T-cell leukemia virus, type 1 (HTLV-1), hepatitis B virus (HBV), or hepatitis C virus (HCV), if allowed by local regulations:

   * Participants with hepatitis B (hepatitis B virus surface antigen [HbsAg] positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid). Participants with HCV with undetectable virus after treatment are eligible. Participants with a prior history of hepatitis B virus are eligible if quantitative polymerase change reaction for hepatitis B virus DNA is negative
   * Participants with human immunodeficiency virus (HIV) infection with acquired immune deficiency syndrome (AIDS) defining illness are not eligible for enrollment; however, participants who have had HIV infection and who have a cluster of differentiation 4 (CD4) + T cell count >350 cells/μL and no history of an AIDS-defining illness are eligible for entry
10. Has an active second malignancy. Note: participants with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or participants with tumors cured with radiotherapy or surgery with low risk of recurrence (e.g., non melanoma skin cancer, histologically confirmed complete excision of carcinoma in situ) are allowed
11. Participants who in the opinion of the Investigator will not be able to adhere to the schedule of assessments and/or may have difficulties complying with the treatment regimen or are unwilling or unable to comply with procedures required in this protocol
12. Known sensitivity to BHV-1530 or any of the excipients in BHV-1530;
13. History of (noninfectious) clinically significant interstitial lung disease (ILD)/pneumonitis that required steroids, active clinically significant ILD/pneumonitis, or suspected clinically significant ILD/pneumonitis that cannot be ruled out by imaging at screening.
14. Requires supplemental oxygen for daily activities
15. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Dose-escalation and Dose-expansion Cohorts: Number of patients with AEs | Through study completion, estimated as an average of 48 months
  Incidence and severity of treatment emergent adverse events (TEAEs), including dose-limiting toxicities (DLTs) and serious adverse events (SAEs)
Dose-confirmation Cohorts: Recommended dose of BHV-1530 for later phase trials | Through study completion, estimated as an average of 48 months
  Incidence and severity of adverse events (AEs) and SAEs, dose reductions during treatment, study discontinuation rates due to TEAEs, and signals of antitumor activity

SECONDARY OUTCOMES:
Dose-escalation and Dose-expansion Cohorts: Clinical Benefit Rate (CBR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-escalation and Dose-expansion Cohorts: Objective Response Rate (ORR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-escalation and Dose-expansion Cohorts: Disease Control Rate (DCR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-escalation and Dose-expansion Cohorts: Time to Response (TTR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-escalation and Dose-expansion Cohorts: Duration of Response (DOR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-escalation and Dose-expansion Cohorts: Progression-free Survival (PFS) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-escalation and Dose-expansion Cohorts: Maximum observed serum concentration (Cmax) | Through study completion, estimated as an average of 48 months
  Serum concentration of BHV-1530, total antibody and TopoIx BHV-0080269
Dose-escalation and Dose-expansion Cohorts: Time of maximum concentration (Tmax) | Through study completion, estimated as an average of 48 months
  Time of maximum concentration of BHV-1530, total antibody and TopoIx BHV-0080269
Dose-escalation and Dose-expansion Cohorts: Elimination half-life (t½) | Through study completion, estimated as an average of 48 months
  Terminal elimination half-life (t½) of BHV-1510, total antibody and TopoIx BHV-0080269
Dose-escalation and Dose-expansion Cohorts: Area Under the Concentration versus time curve (AUC) | Through study completion, estimated as an average of 48 months
  Area under the concentration-time curve from zero to last quantifiable concentration (AUC0-t) and AUC extrapolated to infinity (AUC0-inf) and AUC over the dosing interval (AUCtau)
Dose-escalation and Dose-expansion Cohorts: Trough concentration (Ctrough) | Through study completion, estimated as an average of 48 months
  Trough concentration of BHV-1530, total antibody and TopoIx BHV-0080269
Dose-escalation and Dose-expansion Cohorts: Total body clearance (CL) | Through study completion, estimated as an average of 48 months
  Total body clearance of BHV-1530 and total antibody
Dose-escalation and Dose-expansion Cohorts: Volume of distribution at steady state (Vss) | Through study completion, estimated as an average of 48 months
  Volume of distribution of BHV-1530 and total antibody
Dose-confirmation Cohorts: Objective Response Rate (ORR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-confirmation Cohorts: Disease Control Rate (DCR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-confirmation Cohorts: Time to Response (TTR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-confirmation Cohorts: Duration of Response (DOR) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-confirmation Cohorts: Progression-free Survival (PFS) | Through study completion, estimated as an average of 48 months
  Assessed by RECIST v 1.1
Dose-confirmation Cohorts: Maximum observed serum concentration (Cmax) | Through study completion, estimated as an average of 48 months
  Serum concentration of BHV-1530, total antibody and free payload TopoIx BHV-0080269
Dose-confirmation Cohorts: Time of maximum concentration (Tmax) | Through study completion, estimated as an average of 48 months
  Time of maximum concentration of BHV-1530, total antibody and TopoIx BHV-0080269
Dose-confirmation Cohorts: Elimination half-life (t½) of BHV-1530 | Through study completion, estimated as an average of 48 months
  Terminal elimination half-life (t½) of BHV-1510, total antibody and TopoIx BHV-0080269
Dose-confirmation Cohorts: Area Under the Concentration versus time curve (AUC) | Through study completion, estimated as an average of 48 months
  Area under the concentration-time curve from zero to last quantifiable concentration (AUC0-t) and AUC extrapolated to infinity (AUC0-inf) and AUC over the dosing interval (AUCtau)
Dose-confirmation Cohorts: Trough concentration (Ctrough) | Through study completion, estimated as an average of 48 months
  Trough concentration of BHV-1530, total antibody and TopoIx BHV-0080269
Dose-confirmation Cohorts: Total body clearance (CL) | Through study completion, estimated as an average of 48 months
  Total body clearance of BHV-1530 and total antibody
Dose-confirmation Cohorts: Volume of distribution at steady state (Vss) | Through study completion, estimated as an average of 48 months
  Volume of distribution of BHV-1530 and total antibody

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Site-107, Denver, Colorado
  - Site-108, Lake Mary, Florida
  - Site-110, Detroit, Michigan
  - Site-115, Durham, North Carolina
  - Site-112, Myrtle Beach, South Carolina
  - Site-116, Nashville, Tennessee
  - Site-103, Austin, Texas
  - Site-104, Houston, Texas
  - Site-101, Irving, Texas
  - Site-105, San Antonio, Texas
  - Site-106, West Valley City, Utah
  - Site-102, Fairfax, Virginia